CLINICAL TRIAL: NCT04144335
Title: A Phase 1B Study of N-803 Combined With the Broadly Neutralizing Antibodies VRC07-523LS and PGT121 Plus or Minus haNK Cells for Reduction of HIV Reservoirs
Brief Title: N-803 Combined With the Broadly Neutralizing Antibodies Plus or Minus haNK Cells for HIV
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Contact issues
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007810
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hiv; HIV/AIDS; HIV Infections; AIDS; AIDS and Infections; Aids/Hiv Problem
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Infections | interventions — ALT-803; Broadly Neutralizing Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: N-803 and bNAbs Only (Active Comparator): Group 1 will receive only N-803 and the bNAbs; they will not receive the haNK™ cells
  Interventions: Biological: N-803 and bNAbs
- Group 2: N-803 and bNAbs with haNK™ Cells (Experimental): The protocol for Group 2 will be identical to the one followed by Group 1, except that they will receive haNK™ cells on the same day as each dose of N-803.
  Interventions: Biological: N-803 and bNAbs; Biological: haNK™ Cells

INTERVENTIONS:
Biological: N-803 and bNAbs — Treatment will consist of N-803, VRC07-523LS, PGT121, and haNK, with N-803 given for 3 cycles of 9 weeks/cycle. N-803 will be given every 3 weeks (3 doses/cycle) and bNAbs will be given every 9 weeks.
Biological: haNK™ Cells — Treatment will consist of N-803, VRC07-523LS, PGT121, and haNK, with N-803 given for 3 cycles of 9 weeks/cycle. N-803 will be given every 3 weeks (3 doses/cycle), bNAbs will be given every 9 weeks, and haNK cells administered on the same day as each infusion of N-803.
  Arms: Group 2: N-803 and bNAbs with haNK™ Cells

SUMMARY:
To assess the safety of combination immune therapy in HIV-infected participants whose HIV is controlled with ART, by determining the incidence and severity of adverse events.

DETAILED DESCRIPTION:
This is a phase 1b study to examine the safety, tolerability and efficacy of the combination of 4 immunotherapies for treatment of HIV in participants with controlled HIV viremia and stable CD4 counts on antiretroviral therapy (ART).

The study will be conducted in two separate phases using two distinct to groups of participants where each group will have 10 individuals enrolled.

Treatment will consist of N-803, VRC07-523LS, PGT121, and haNK, with N-803 given for 3 cycles of 9 weeks/cycle. N-803 will be given every 3 weeks (3 doses/cycle), bNAbs will be given every 9 weeks, and haNK cells administered on the same day as each infusion of N-803. Total study duration will be 27 weeks.

Group 1 will receive only N-803 and the bNAbs; they will not receive the haNK™ cells. When 2 participants are enrolled and on active treatment for one month in Group 1, the Safety Monitoring Committee will review all data and if there are no safety concerns raised in the data recorded from administration of the interventions to those participants, Group 1 will continue. When Group 1 is complete, the SMC will again review all data before Group 2 can proceed with enrollment. The protocol for Group 2 will be identical to the one followed by Group 1, except that they will receive haNK™ cells at 2 × 109 cells/dose IV on the same day as each dose of N-803.

Optional tissue biopsies (lymph node and colonoscopy to collect gut-associated lymphoid tissue (GALT)) will occur at baseline and again 9 weeks after the last infusion of bNAbs. We aim to perform biopsies on least 8 out of 10 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* On continuous antiretroviral therapy for > 12 months without any interruptions of greater than 14 consecutive days in the last 12 months
* Screening plasma HIV RNA levels < 20 copies/mL on all available determinations in past 12 months (isolated single values ≥ 20 but < 200 copies/mL will be allowed if they were preceded and followed by viral load determinations < 20 copies/mL)
* Screening CD4+ T-cell count ≥ 400 cells/mm3

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Active or recent malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months; minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) are not exclusionary
* Chronic liver disease defined as Class B and C on the Child-Pugh scale
* Active and poorly controlled atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 ACC/AHA guidelines, including a previous diagnosis of any of the following: (a) acute myocardial infarction, (b) acute coronary syndromes, (c) stable or unstable angina, (d) coronary or other arterial revascularization, (e) stroke, (f) transient ischemic attack (TIA), or (g) peripheral arterial disease grade IIa or greater
* History of AIDS-defining illness within the past 5 years
* History of potential immune-mediated medical conditions requiring concomitant treatment with immunomodulatory drugs, and/or exposure to any immunomodulatory drug in the 4 weeks prior to study enrollment
* Exposure to any experimental therapies within 90 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of Adverse Events Grades 3, 4, 5 | 27 weeks
  Number of serious adverse events (SAEs) graded 3 (severe pain; interferes with oral intake), 4 (life-threatening consequences; urgent intervention needed), and 5 (death) experienced in the haNK cell group compared to the group receiving no haNK cells. Lower number of SAEs indicated greater treatment safety.

SECONDARY OUTCOMES:
Reduction of HIV Reservoir in PBMCs | 27 weeks
  HIV RNA in peripheral blood mononuclear cells (PBMCs) will be quantified using next gen sequencing. Percent reduction in HIV RNA reservoirs in these cells will be compared between groups. Greater percent reduction in viral reservoirs in haNK cell group indicates greater efficacy of haNK cell therapy compared to no haNK cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Schacker, MD, Principal Investigator — Medical School, University of Minnesota
Locations (3):
- United States (3):
  - University of California, San Francisco, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No